CLINICAL TRIAL: NCT03816163
Title: A Phase 2, Open-Label, Randomized Study to Assess the Efficacy and Safety of Zolbetuximab (IMAB362) in Combination With Nab-Paclitaxel and Gemcitabine (Nab-P + GEM) as First Line Treatment in Subjects With Claudin 18.2 (CLDN18.2) Positive, Metastatic Pancreatic Adenocarcinoma
Brief Title: A Study of Zolbetuximab (IMAB362) in Adults With Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8951-CL-5201; 2018-002551-15 (EudraCT Number); CTR20220914 (Registry Identifier: ChinaDrugTrials.org.cn); 2024-510985-17-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT06048081 (Available)
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer; Metastatic Pancreatic Cancer; Metastatic Pancreatic Adenocarcinoma
Keywords: metastatic pancreatic cancer; IMAB362; nab-paclitaxel; gemcitabine; zolbetuximab; metastatic pancreatic adenocarcinoma; pancreatic cancer; CLDN 18.2
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — zolbetuximab; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- zolbetuximab +nab-paclitaxel + gemcitabine (Experimental): Participants will be treated with zolbetuximab in combination with nab-paclitaxel and gemcitabine for the phase 1 portion of the study to establish the recommended dose of zolbetuximab for the phase 2 portion. In the phase 2 portion, the participants will be treated with zolbetuximab at dose determined by the phase 1 portion of the study in combination with nab-paclitaxel and gemcitabine. Participants will be treated on continuous cycles until they no longer derive clinical benefit in the judgment of the treating physician, have unacceptable toxicity, undergo hematopoietic stem cell transplantation (HSCT), or meet one of the discontinuation criteria; whichever occurs first.
  Interventions: Drug: zolbetuximab; Drug: nab-paclitaxel; Drug: gemcitabine
- nab-paclitaxel + gemcitabine (Active Comparator): Participants will be treated with nab-paclitaxel and gemcitabine. Participants will be treated on continuous cycles until they no longer derive clinical benefit in the judgment of the treating physician, have unacceptable toxicity, undergo hematopoietic stem cell transplantation (HSCT), or meet one of the discontinuation criteria; whichever occurs first.
  Interventions: Drug: nab-paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: zolbetuximab — Administered as an intravenous infusion.
  Other Names: IMAB362
  Arms: zolbetuximab +nab-paclitaxel + gemcitabine
Drug: nab-paclitaxel — Administered as an intravenous infusion
Drug: gemcitabine — Administered as an intravenous infusion

SUMMARY:
Zolbetuximab is being studied as a treatment for people with pancreatic cancer. Most people with pancreatic cancer have a protein called Claudin 18.2 (CLDN18.2) in their tumor. Zolbetuximab is thought to work by attaching to CLDN 18.2 in their tumor. This switches on the body's immune system to attack the tumor. Zolbetuximab is a potential treatment for people with pancreatic cancer.

There is an unmet medical need to treat people with pancreatic cancer. This study will help find the dose of zolbetuximab to be used with chemotherapy and provide more information on this treatment in adults with metastatic pancreatic cancer. The study is currently ongoing globally. People in this study will be treated with either zolbetuximab and chemotherapy or chemotherapy by itself.

The study's main aims are to find a suitable dose of zolbetuximab to be used with chemotherapy in the second part of this study, to check if zolbetuximab and chemotherapy compared to chemotherapy by itself can improve the survival of people with pancreatic cancer, and to check the safety of zolbetuximab when given with chemotherapy and how well people cope with medical problems during the study.

Adults with metastatic pancreatic cancer can take part. Their cancer is metastatic, has the CLDN18.2 marker in a tumor sample and has not previously been treated with chemotherapy. Metastatic means the cancer has spread to other parts of the body. People cannot take part are if they have recently had radiotherapy and have not recovered, need to take medicines to suppress their immune system, have history of nervous system metastases from their pancreatic cancer, or they have other active cancers that need treatment. People who have a specific heart condition or infections also cannot take part.

This study will be in 2 parts. Part 1 is called the Safety Lead-in Phase. Groups of people will receive 1 of 2 different doses of zolbetuximab: a lower dose or a higher dose, both together with chemotherapy. A medical expert panel will check the results and decide the dose to use in Part 2.

Part 2 is called the Randomization Phase. People will be put in 1 of 2 groups by chance and will be given different treatments either zolbetuximab and chemotherapy or chemotherapy by itself. The chance of receiving zolbetuximab and chemotherapy is twice as high as receiving chemotherapy by itself. In both parts of the study, zolbetuximab and chemotherapy or chemotherapy by itself will be given through a vein. This is called an infusion. Each treatment cycle is 4 weeks (28 days) long and people will have either 2 infusions of zolbetuximab and 3 infusions of chemotherapy or 3 infusions of chemotherapy by itself during each treatment cycle. People will visit the clinic on certain days during their treatment. The study doctors will check for any medical problems from zolbetuximab. Also, people in the study will have a health check including blood tests. On some visits they will also have scans to check for any changes in their cancer. Tumor samples will be taken before treatment if a previous sample is not available. People will have the option of giving a tumor sample after treatment has finished. People will visit the clinic after they stop treatment. They will be asked about any medical problems and will have a health check including blood tests. The number of visits and checks done at each visit will depend on the health of each person and whether they completed their treatment or not.

DETAILED DESCRIPTION:
This study will have a safety lead in phase and a randomization phase.

ELIGIBILITY:
Inclusion Criteria:

* A female subject is eligible to participate if she is not pregnant or lactating and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 6 months after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* A male subject with female partner(s) of child-bearing potential must agree to use contraception during the treatment period and for at least 6 months after the final study drug administration.
* A male subject must not donate sperm during the treatment period and for at least 6 months after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 6 months after the final study drug administration.
* Subject agrees not to participate in other interventional studies while receiving study drug in present study.
* Subject has histologically or cytologically confirmed adenocarcinoma of pancreas.
* Subjects must have metastatic pancreatic adenocarcinoma that has not been previously treated with chemotherapy.

  * Prior treatment with fluorouracil (5-FU) or GEM administered as a radiation sensitizer during and up to 4 weeks after radiation therapy is allowed
  * If a subject received adjuvant therapy, tumor recurrence or disease progression must have occurred at least 6 months after completing the last dose of the adjuvant therapy.
  * Subjects whose disease progressed on prior treatment with Nab-P and GEM are not eligible.
* Subject has a measurable lesion(s) on at least 1 metastatic site based on RECIST 1.1 within 28 days prior to randomization. For subjects with only 1 measurable lesion and prior radiotherapy, the lesion must be outside the field of prior radiotherapy or must have documented progression following radiation therapy.
* Subject's tumor sample has CLDN18.2 expression in ≥ 75% of tumor cells demonstrating moderate to strong membranous staining as determined by central immunohistochemistry (IHC) testing
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subject has predicted life expectancy ≥ 12 weeks.
* Subject must meet all of the following criteria based on the laboratory tests that will be collected within 14 days prior to randomization. In case of multiple laboratory data within this period, the most recent data should be used.

  * Hemoglobin ≥ 9 g/dl (no transfusion within 14 days of start of study treatment)
  * Absolute neutrophil count ≥ 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Albumin ≥ 2.5 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN without liver metastases (≤ 5 x ULN if liver metastases are present)
  * Estimated creatinine clearance ≥ 30 mL/min
  * Prothrombin time/international normalized ratio (INR) and partial thromboplastin time ≤ 1.5 x ULN (except for subjects receiving anticoagulation therapy)

Exclusion Criteria:

* Subject has received other investigational treatment within 28 days prior to randomization.
* Subject has received radiotherapy for metastatic pancreatic adenocarcinoma ≤ 14 days prior to randomization and has not recovered from any related toxicity.
* Subject has received systemic immunosuppressive therapy, including systemic corticosteroids within 14 days prior to randomization. Subject using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone), receiving a single dose of systemic corticosteroids or receiving systemic corticosteroids as premedication for radiologic imaging contrast use are allowed.
* Subject has prior severe allergic reaction or intolerance to known ingredients of zolbetuximab or other monoclonal antibody, including humanized or chimeric antibodies.
* Subject has known immediate or delayed hypersensitivity, intolerance or contraindication to any component of study treatment.
* Subject has a known history of a positive test for human immunodeficiency virus infection or known active hepatitis B (positive HBs antigen [Ag]) or hepatitis C infection. NOTE: Screening for these infections should be conducted per local requirements.

  1. For subjects who are negative for HBs Ag, but hepatitis B core antibody positive, a hepatitis B virus DNA test will be performed and if positive, the subject will be excluded.
  2. Subjects with positive hepatitis C serology but negative hepatitis C virus RNA test results are eligible.
  3. Subjects treated for hepatitis C with undetectable viral load results are eligible.
* Subject has a history of interstitial pneumonia or pulmonary fibrosis.
* Subject has pleural effusion or ascites ≥ Grade 3.
* Subject has an active autoimmune disease that has required systemic treatment in the past 3 months prior to randomization.
* Subject has active infection requiring systemic therapy that has not completely resolved per investigator judgment within 7 days prior to randomization.
* Subject has significant cardiovascular disease, including:

  * Congestive heart failure (defined as New York Heart Association Class III or IV), myocardial infarction, unstable angina, coronary angioplasty, coronary stenting, coronary artery bypass graft, cerebrovascular accident or hypertensive crisis within 6 months prior to randomization;
  * History of clinically significant ventricular arrhythmias (i.e., sustained ventricular tachycardia, ventricular fibrillation or Torsades de Pointes);
  * QTc interval > 450 msec for male subjects; QTc interval > 470 msec for female subjects;
  * Cardiac arrhythmias requiring anti-arrhythmic medications (Subjects with rate controlled atrial fibrillation for > 1 month prior to randomization.)
* Subject has a history of central nervous system metastases and/or carcinomatous meningitis from pancreatic adenocarcinoma.
* Subject has known peripheral sensory neuropathy ≥ Grade 2 unless the absence of deep tendon reflexes is the sole neurological abnormality.
* Subject has had a major surgical procedure ≤ 28 days prior to randomization.
* Subject without complete recovery from a major surgical procedure ≤ 14 days prior to randomization.
* Psychiatric illness or social situations that would preclude study compliance.
* Subject has another malignancy for which treatment is required.
* Subject has any concurrent disease, infection or co-morbid condition that interferes with the ability of the subject to participate in the study, which places the subject at undue risk or complicates the interpretation of data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) - (safety lead in) | Up to 28 days
  Incidence of dose limiting toxicities.
Overall Survival (OS) | Up to 65 months
  OS is defined as the time from the date of randomization until the date of death from any cause.
Safety assessed by Adverse Events (AEs) | Up to 65 months
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Safety assessed by incidence of serious adverse events (SAE) | Up to 65 months
  Adverse Event (AE) is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event.
Safety assessed by incidence of treatment emergent adverse events (TEAE) | Up to 65 months
  Treatment Emergent Adverse Event (TEAE) is defined as any AE which starts, or worsens, after the first dose of study drug through 30 days after the last dose of study drug.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 65 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and /or adverse events (AEs) | Up to 65 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiograms (ECG) abnormalities and or adverse events | Up to 65 months
  12-lead ECGs will be recorded. Prior to the ECG, participants should rest in supine position for 10 minutes. ECGs will be read and assessed locally.
Number of participants with Eastern Cooperative Oncology Group (ECOG) performance status abnormalities and or adverse events | Up to 65 months
  Number of participants with potentially clinically significant ECOG performance status values. ECOG grades 0-5, where 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair and 5 = Dead.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 65 months
  PFS is defined as the time from the date of randomization until the date of radiological progressive disease (PD) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 by investigator evaluation or death from any cause, whichever is earliest.
Objective Response Rate (ORR) | Up to 65 months
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by investigator evaluation per RECIST 1.1.
Number of anti-drug antibody (ADA) Positive Participants | Up to 65 months
  Immunogenicity will be measured by the number of participants that are ADA positive.
Disease Control Rate (DCR) | Up to 65 months
  DCR is defined as the proportion of participants who have best overall response of stable disease, complete response (CR) or partial response (PR) as assessed by investigator evaluation per RECIST 1.1
Duration Of Response (DOR) | Up to 65 months
  DOR is defined as the time from the date of the first response (CR/PR) until the date of progressive disease as assessed by investigator evaluation per RECIST 1.1 or date of death from any cause, whichever is earliest.
Change in CA (Cancer Antigen) 19-9 | Baseline up to 65 months
  Change from baseline in serum CA19-9 will be assessed.
PK of zolbetuximab: Concentration Immediately Prior to Dosing (Ctrough) | Up to 65 months
  Ctrough will be derived from the PK serum samples collected.
PK of Nab-P: Area Under the Concentration-time Curve from the Time of Dosing Extrapolated to Time Infinity (AUCinf) | Up to 30 days
  AUCinf will be derived from the PK plasma samples collected.
PK of Nab-P: Area Under the Concentration-time Curve from the Time of Dosing Until the Last Measurable Concentration (AUClast) | Up to 30 days
  AUClast will be derived from the PK plasma samples collected.
PK of Nab-P: Maximum Concentration (Cmax) | Up to 30 days
  Cmax will be derived from the PK plasma samples collected.
PK of Nab-P: Time of Maximum Concentration (Tmax) | Up to 30 days
  Tmax will be derived from the PK plasma samples collected.
PK of Nab-P: Terminal Elimination Half-life (T1/2) | Up to 30 days
  T1/2 will be derived from the PK plasma samples collected.
PK of Nab-P: Clearance (CL) | Up to 30 days
  CL will be derived from the PK plasma samples collected.
PK of Nab-P: Volume of Distribution During the Terminal Phase (Vz) | Up to 30 days
  Vz will be derived from the PK plasma samples collected.
PK of gemcitabine: Area Under the Concentration-time Curve from the Time of Dosing Extrapolated to Time Infinity (AUCinf) | Up to 30 days
  AUCinf will be derived from the PK plasma samples collected.
PK of gemcitabine: Area Under the Concentration-time Curve from the Time of Dosing Until the Last Measurable Concentration (AUClast) | Up to 30 days
  AUClast will be derived from the PK plasma samples collected.
PK of gemcitabine: Maximum Concentration (Cmax) | Up to 30 days
  Cmax will be derived from the PK plasma samples collected.
PK of gemcitabine: Time of Maximum Concentration (Tmax) | Up to 30 days
  Tmax will be derived from the PK plasma samples collected.
PK of gemcitabine: Terminal Elimination Half-life (T1/2) | Up to 30 days
  T1/2 will be derived from the PK plasma samples collected.
PK of gemcitabine: Clearance (CL) | Up to 30 days
  CL will be derived from the PK plasma samples collected.
PK of gemcitabine: Volume of Distribution During the Terminal Phase (Vz) | Up to 30 days
  Vz will be derived from the PK plasma samples collected.
Health Related Quality of Life (HRQoL) measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core Questionnaire (EORTC-QLQ-C30) | Up to 65 months
  The EORTC-QLQ-C30 is a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." For functional scales, higher scores indicate better functioning, while for symptom scales/items, higher scores indicate worse symptoms.
Health Related Quality of Life (HRQoL) measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Pancreatic Cancer Module (EORTC-QLQ-PAN-26) | Up to 65 months
  EORTC-QLQ-PAN26 is a 26-item questionnaire that evaluates pancreatic cancer-specific symptoms such as pain, dietary changes, jaundice, altered bowel habits, and emotional problems. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." For symptom scales/items, higher scores indicate worse symptoms.
Health Related Quality of Life (HRQoL) measured by the EuroQOL Five Dimensions Questionnaire 5L (EQ-5D-5L) | Up to 65 months
  The EQ-5D-5L is a standardized instrument for use as a measure of health outcome consisting of 6 items that cover 5 main domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a general visual analog scale for health status.
  Each domain comprises 5 severity levels (no problems, slight problems, moderate problems, severe problems, extreme problems). The general visual analog scale records the respondent's self-rated health status on a vertical graduated (0 = the worst health a participant can imagine to 100 = the best health a participant can imagine) visual analogue scale. Responses to the 5 items will also be converted to a weighted health state index (utility score) based on values derived from general population samples.
Health Related Quality of Life (HRQoL) measured by the Patient Global Impression of Change (PGIC) scale | Up to 65 months
  The PGIC is a single-item questionnaire that asks participants to provide the overall self-assessment of change in their disease on a 7-point scale ranging from "very much worse" to "very much better" as compared to the participant starting the study treatment. Only PGIC questions assessing pain and overall status will be collected.
Health Related Quality of Life (HRQoL) measured by the Patient Global Impression of Severity (PGIS) Scale | Up to 65 months
  The PGIS is a single-item questionnaire that asks participants to provide the overall self-assessment of their disease severity on a 4-point scale for the past week, with 1 as "None" and 4 as "Severe". Only PGIS questions assessing pain and overall status will be collected.
Time to Improvement of pancreatic pain as measured by Quality-of-Life Questionnaire - Core Questionnaire (QLQ-C30) | Up to 65 months
  The QLQ-C30 is a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." For functional scales, higher scores indicate better functioning, while for symptom scales/items, higher scores indicate worse symptoms.
Time to worsening of global health status (GHS)/quality of life (QoL) as measured by QLQ-C30 | Up to 65 months
  The QLQ-C30 is a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." For functional scales, higher scores indicate better functioning, while for symptom scales/items, higher scores indicate worse symptoms.
Time to Improvement of pancreatic pain as measured by Quality of Life Questionnaire - Pancreatic Cancer Module 26 (QLQ-PAN26) | Up to 65 months
  EORTC-QLQ-PAN26 is a 26-item questionnaire that evaluates pancreatic cancer-specific symptoms such as pain, dietary changes, jaundice, altered bowel habits, and emotional problems. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." For symptom scales/items, higher scores indicate worse symptoms.
Time to worsening of GHS/QoL as measured by QLQ-PAN26 | Up to 65 months
  EORTC-QLQ-PAN26 is a 26-item questionnaire that evaluates pancreatic cancer-specific symptoms such as pain, dietary changes, jaundice, altered bowel habits, and emotional problems. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." For symptom scales/items, higher scores indicate worse symptoms.
Time to Improvement of pancreatic pain as measured by PGIS | Up to 65 months
  The PGIS is a single-item questionnaire that asks participants to provide the overall self-assessment of their disease severity on a 4-point scale for the past week, with 1 as "None" and 4 as "Severe". Only PGIS questions assessing pain and overall status will be collected.
Time to worsening of GHS/QoL as measured by PGIS | Up to 65 months
  The PGIS is a single-item questionnaire that asks participants to provide the overall self-assessment of their disease severity on a 4-point scale for the past week, with 1 as "None" and 4 as "Severe". Only PGIS questions assessing pain and overall status will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (136):
- United States (25):
  - St. Joseph Heritage Medical Group, Fullerton, California
  - TOI Clinical research, Whittier, California
  - Midstate Medical Center, Meriden, Connecticut
  - Lynn Cancer Institute, Boca Raton, Florida
  - Baptist Health, Miami, Florida
  - Cancer Treatment Centers of Atlanta, Newnan, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Norton Cancer Institute (NCI), Louisville, Kentucky
  - Ochsner Health System, New Orleans, Louisiana
  - David C Pratt Cancer Center, Creve Coeur, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health Cancer Institute, Lake Success, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - Houston Methodist Hospital, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - MultiCare Regional Cancer Center - Gig Harbor, Gig Harbor, Washington
  - Vista Oncology, Olympia, Washington
  - Virginia Mason, Seattle, Washington
- Australia (4):
  - Site AU61008, Gosford, New South Wales
  - Site AU61007, Wollongong, New South Wales
  - Site AU61005, Fitzroy, Victoria
  - Site AU61006, Warrnambool, Victoria
- Brazil (6):
  - Site BR55012, Porto Alegre, Rio Grande do Sul
  - Site BR55009, Centro Passo Fundo
  - Site BR55008, Rio Grande
  - Site BR55004, Santa Catarina
  - Site BR55010, São Paulo
  - Site BR55011, São Paulo
- China (23):
  - Site CN86001, Beijing
  - Site CN86008, Beijing
  - Site CN86014, Beijing
  - Site CN86026, Changchun
  - Site CN86009, Chongqing
  - Site CN86004, Guangdong
  - Site CN86020, Guangdong
  - Site CN86016, Guangzhou
  - Site CN86012, Harbin
  - Site CN86002, Hubei
  - Site CN86005, Jiangsu
  - Site CN86011, Jiangsu
  - Site CN86025, Jiangsu
  - Site CN86023, Shandong
  - Site CN86006, Shanghai
  - Site CN86013, Shanghai
  - Site CN86019, Shanghai
  - Site CN86007, Tianjin
  - Site CN86022, Xinjiang
  - Site CN86024, Yanxi
  - Site CN86003, Zhejiang
  - Site CN86018, Zhejiang
  - Site CN86010, Zhengzhou
- France (19):
  - Site FR33008, Besançon, Besancon Cedex
  - Site FR33010, Brest, Brest Cedex
  - Site FR33015, Caen, Cedex 5
  - Site FR33006, Chambray, Cedex 9
  - Site FR33012, Herblain, Herblain Cedex
  - Site FR33016, La Chaussée-Saint-Victor, Loir-et-Cher
  - Site FR33009, Nancy, Nancy Cedex
  - Site FR33017, Rouen, Normandy
  - Site FR33003, Aquitaine, Pessac
  - Site FR33013, Villejuif, Villejuif Cedex
  - Site FR33001, Bayonne
  - Site FR33018, Bordeaux
  - Site FR33002, Grenoble
  - Site FR33019, La Roche-sur-Yon
  - Site FR33021, Nice
  - Site FR33023, Pierre-Bénite
  - Site FR33014, Plérin
  - Site FR33005, Pringy
  - Site FR33007, Strasbourg
- Site IR35301, Elm Park, Dublin, Ireland
- Italy (7):
  - Site IT39006, Rozzano, Milan
  - Site IT39004, Candiolo, Torino
  - Site IT39002, Cremona
  - Site IT39010, Lombardia
  - Site IT39003, Milan
  - Site IT39014, Toscana
  - Site IT39008, Veneto
- Japan (14):
  - Site JP81007, Nagoya, Aichi-ken
  - Site JP81001, Kashiwa, Chiba
  - Site JP81005, Sapporo, Hokkaido
  - Site JP81006, Yokohama, Kanagawa
  - Site JP81003, Kashihara, Nara
  - Site JP81011, Bunkyo-ku, Tokyo
  - Site JP81012, Chuo-ku, Tokyo
  - Site JP81014, Koto-ku, Tokyo
  - Site JP81013, Mitaka, Tokyo
  - Site JP81002, Shinjuku-ku, Tokyo
  - Site JP81015, Ube, Yamaguchi
  - Site JP81004, Fukuoka
  - Site JP81010, Osaka
  - Site JP81009, Wakayama
- Mexico (3):
  - Site MX52004, Distrito Federal
  - Site MX52003, San Luis Potosí City
  - Site MX52005, Veracruz
- South Korea (10):
  - Site KR82005, Seongnam-si, Gyeonggi-do
  - Site KR82008, Suwon, Gyeonggi-do
  - Site KR82010, Daegu
  - Site KR82009, Gyeonggi-do
  - Site KR82001, Seoul
  - Site KR82003, Seoul
  - Site KR82004, Seoul
  - Site KR82007, Seoul
  - Site KR82002, Seoul
  - Site KR82006, Seoul
- Spain (15):
  - Site ES34004, Llobregat, Barcelona
  - Site ES34003, Pamplona, Navarre
  - Site ES34010, Barcelona
  - Site ES34013, Barcelona
  - Site ES34007, Barcelona
  - Site ES34018, Barcelona
  - Site ES34021, Barcelona
  - Site ES34014, Cáceres
  - Site ES34022, Córdoba
  - Site ES34005, Lleida
  - Site ES34015, Madrid
  - Site ES34006, Madrid
  - Site ES34009, Madrid
  - Site ES34026, Málaga
  - Site ES34017, Santiago de Compostela
- Taiwan (4):
  - Site TW88608, New Taipei City
  - Site TW88602, Taichung
  - Site TW88601, Taipei
  - Site TW88609, Taipei
- Turkey (Türkiye) (5):
  - Site TR90004, Ankara
  - Site TR90006, Ankara
  - Site TR90003, Diyarbakır
  - Site TR90002, Istanbul
  - Site TR90001, Konya

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/